CLINICAL TRIAL: NCT06985927
Title: Self-Concept and Autobiographical Memory in the Care of Patients With Alcohol Use Disorder
Brief Title: Self-Concept and Autobiographical Memory in Alcohol Use Disorder
Acronym: CoSMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PO25057*
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorders; Self-Concept; Autobiographical Memory; Psychotherapeutic Care
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of two or more groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Self-Concept Group (Experimental)
  Interventions: Behavioral: psychotherapeutic sessions

INTERVENTIONS:
Behavioral: psychotherapeutic sessions — Analysis of effect of psychotherapeutic sessions based on self-concept and autobiographical memory on alcohol addiction
  Arms: Self-Concept Group

SUMMARY:
This study has two objectives. First, to evaluate the effectiveness of psychotherapy sessions based on self-concept and autobiographical memory in patients suffering from alcohol use disorders (AUD). Second, investigate the relationship between drinking identity and AUD. These objectives will be investigated according to a longitudinal design.

In this study, the drinking identity is evaluated on its implicit dimension and on its explicit dimension. Levels of alcohol use and dependence are assessed by the amount and frequency of drinking, the duration of abstinence, and the intensity of AUD symptoms. These assessments consist three visits: on the day of inclusion, then at three months and six months after the first visit. The psychotherapy sessions consist of four individual sessions. They are inspired by the Social Identity Mapping in Addiction Recovery (SIM-AR) by Beckwith et al. (2019), combined with autobiographical reasoning exercises.

Patients with an AUD, participants in the study, are recruited from the addiction department of the Etablissement Public de Santé Mentale de la Marne. To investigate the effects of individual psychotherapy sessions, two groups of patients are constituted randomly. The first group will have four psychotherapy sessions between the first visit and the second vist. The second group will not follow psychotherapy sessions but will benefit from the usual addiction treatments.

The first hypothesis is that patients who have completed the psychotherapy sessions will have lower alcohol consumption (frequency, quantities, peaks) and symptoms of AUD (cravings, drinking refusal self-efficacy and feeling of recovery) than those who have not benefited from the program.

The second hypothesis is that implicit and explicit levels of drinking identity will predict alcohol consumption (frequencies, quantities, peaks) and symptoms of dependence (cravings, drinking refusal self-efficacy and feeling of recovery) for all participants.

DETAILED DESCRIPTION:
BACKGROUND Surveys on the proportion of deaths attributable to alcohol consumption consider this practice to be the second cause of avoidable mortality in France. The first victims of alcohol consumption are patients with Alcohol Use Disorder (AUD). This chronic and complex pathology requires treatment that takes into account many factors of biological, psychological and social origin. From this perspective, one of the factors highlighted in the understanding of drinking behavior is the drinking identity. Drinking identity is the integration, more or less conscious, of alcohol as part of one's self-concept. It works in two dimensions, based on the dual-process model of Strack and Deutsch: an implicit dimension and an explicit dimension. A recent meta-analysis showed that, in the general population, the drinking identity is a robust predictor of drinking behaviors and the problems associated. Thus, the drinking identity appears to be a particularly relevant field of research and intervention within the framework of the AUD. To help patients with AUD to change their drinking identity, this study proposes to evaluate the interest of psychotherapeutic workshops focused on Autobiographical Memory (AM) and self-concept. This form of memory stores all of an individual's autobiographical information and memories. AM has the elements that help individuals to build a coherent image of themselves and to update their self-concept. Thus, AM could be a therapeutic lever towards drinking identity.

STUDY PROCEDURES This longitudinal study has two aims. Firs aims is to analyze the therapeutic effectiveness of psychotherapy sessions based on self-concept and AM for patients with alcohol use disorder. Indeed, the management of AUD has a moderate effectiveness. The search for new tools and therapeutic axes is crucial. The link between drinking identity and alcohol consumption was observed only in a general population, so, the second aim of this study is to observe in people with AUD, the link between the level of drinking identity, alcohol consumption and the level of alcohol dependence.

Plan: 60 patients with AUD will be recruited within the addiction unit of the Etablissement Public de Santé Mentale de la Marne (France). In order to investigate the effects of psychotherapeutic sessions and the relationship between the drinking identity and AUD. This study will follow a longitudinal model. All sixty participants will have three evaluation times (visits): a first evaluation and inclusion visit, a second evaluation visit 3 months later and a third evaluation visit 6 months after the first visit. During these visits, the levels of alcohol consumption and symptoms of dependence are assessed as well as the level of drinking identity.

In addition, to observe the effects of individual psychotherapy sessions, two groups of patients will be constituted randomly (each group is composed of 30 participants). The first group will carries out four psychotherapeutic sessions focused on AM and the self-concept.

Measures For the assessment of alcohol consumption and AUD, several measures are used. For alcohol consumption, the frequency, quantities and peaks of consumption are recorded. For AUD, several dimensions are evaluated: cravings, drinking refusal self-efficacy and feeling of recovery.

Explicit drinking identity is the identity integration of alcohol accessible to consciousness giving during introspection: "Alcohol is part of who I am". Conversely, implicit drinking identity is an unconscious and rapid cognitive process forming one of the elements of the network constituting the "self". And whose link between the self and this representation would be more or less important. The evaluation of the explicit drinking identity will be made through self-questionnaires. Conversely, the implicit drinking identity will be evaluated with computer task: implicit association test.

Finally, other measures are carried out, in particular to observe the link between drinking identity and AM as well as the effect of psychotherapeutic workshops such as: self-defining memory task or self-esteem.

Hypotheses:

The first hypothesis is that patients who will have completed the psychotherapy sessions will have lower alcohol consumption (frequency, quantities, peaks) and lower symptoms of AUD (cravings, drinking refusal self-efficacy and feeling of recovery) than those who have not benefited from the program.

The second hypothesis is that implicit and explicit levels of drinking identity will predict alcohol consumption (frequencies, quantities, peaks) and symptoms of dependence (cravings, drinking refusal self-efficacy and feeling of recovery) for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 24 years old, men or women
* Having a diagnosis of alcohol use disorder according to DSM-5 criteria
* Being a native French speaker
* Patients enrolled in the national healthcare insurance program
* Consenting to participate to the study

Exclusion Criteria:

* A diagnosis of current non-stabilized psychiatric disorders according to DSM-5 criteria
* The presence of another substance use disorder, except for tobacco dependence
* The presence of any intellectual disability, of pervasive developmental disorders
* The presence of any neurological disorder or any other disorder affecting the central nervous system including neurological complications of alcoholism
* A sensorial impairment uncorrected (visual and/or hearing)

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Severity of alcohol use disorder | Day 0, to 3 months, to 6 months
  The Alcohol Use Disorder Inventory Test (AUDIT). The AUDIT is self-administered questionnaire consists of 10 items designed to identify the risk of the presence of an alcohol use disorder with or without dependence. Items 1 to 6 assess the presence of an alcohol use disorder, and items 7 to 10 assess problems associated with the participant's drinking pattern

SECONDARY OUTCOMES:
Craving | Day 0, to 3 months, to 6 months
  Evaluated through Obsessive Compulsive Drinking Scale (OCDS). The OCDS is 12-item self-questionnaire assesses obsessive thoughts and compulsive cravings for alcohol
Drinking refusal self-efficacy | Day 0, to 3 months, to 6 months
  Drinking Refusal Self-Efficacy Questionnaire-Revised (DRSEQ-R) It consists of 19 items in the form of first-person statements, positioned on a 6-point Likert scale. It assesses participants' beliefs about their ability to resist drinking in certain situations on three dimensions: social pressure, emotional relief and opportunistic drinking

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France